CLINICAL TRIAL: NCT01786902
Title: Open, Multi-Center, Controlled, Randomized Phase III Clinical Trial to Evaluate the Efficacy and Safety of DA-3002(Recombinant Humn Growth Hormone)Treatment in Children With Idiopathic Short Stature
Brief Title: Efficacy and Safety of DA-3002 in Children With Idiopathic Short Stature
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA3002_ISS_III
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Idiopathic Short Stature
Keywords: growth hormone
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA-3002 Treatment group (Experimental): 1.11 IU(0.37mg)/kg bodyweight of DA-3002 per week given by subcutaneous injections (six or seven times per week)
  Interventions: Drug: DA-3002
- Non-treatment control group (No Intervention): Height be measured with no treatment

INTERVENTIONS:
Drug: DA-3002
  Other Names: Recombinant Human Growth Hormone
  Arms: DA-3002 Treatment group

SUMMARY:
Growth hormone therapy will improve the height of idiopathic short statured children. DA-3002(Recombinant Human Growth hormone)treated group for 26 weeks, will be compared to non-treatment group in efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Chronological Age ≥ 4
* Bone Age <11 (for girls) and <13 (for boys)
* Height <3rd percentile for age
* normal thyroid function

Exclusion Criteria:

* endocrine and/or metabolic disorders
* growth failure caused by other disorders
* previous use of drugs that could interfere with Growth Hormone treatment

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanwook Yoo, MD, Principal Investigator — Asan Medical Center; Byungkyu Suh, MD, Study Director — Seoul St. Mary's Hospital; Cheolwoo Ko, MD, Study Director — Kyungpook National University Hospital; Keehyoung Lee, MD, Study Director — Korea University Anam Hospitial; Dongkyu Jin, MD, Study Director — Samsung Medical Center; Choongho Shin, MD, Study Director — Seoul National University Hospital; Jinsoon Hwang, MD, Study Director — Aju University Hospital; Hoseong Kim, MD, Study Director — Severance Children's Hospital Yonsei University; Wooyoung Jeong, MD, Study Director — Pusan University Hospital; Chanjong Kim, MD, Study Director — Chonnam National University Hospital; Heonsuk Han, MD, Study Director — Chungbuk National University Hospital

RESULTS

PARTICIPANT FLOW:
Groups:
- DA-3002 Treatment Group: 1.11 IU(0.37mg)/kg bodyweight of DA-3002 per week given by subcutaneous injections (six or seven times per week)
  DA-3002
Period: Overall Study
Arm/Group | DA-3002 Treatment Group | Non-treatment Control Group
Started | 36 | 34
Completed | 32 | 31
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DA-3002 Treatment Group | Non-treatment Control Group | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.75 (1.79) | 7.17 (2.34) | 6.96 (2.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 22 | 17 | 39
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Annualized Height Velocity(cm/Year) After 26 Weeks
Description: Height Velocity calculated with height measured at Baseline and after 26 weeks was converted to annual growth rate.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | DA-3002 Treatment Group | Non-treatment Control Group
Number analyzed (Participants) | 36 | 32
cm/year | 10.68 (1.95) | 5.72 (1.72)

2. Secondary Outcome: Changes in Height Standard Deviation Score After 26 Weeks
Description: The Height Standard Deviation Score was calculated as height minus reference mean height divided by the standard deviation of the reference mean height, both given by a reference growth table for the corresponding chronological age at the height measurement. Greater Height Standard Deviation Score indicates greater height.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DA-3002 Treatment Group | Non-treatment Control Group
Number analyzed (Participants) | 36 | 32
ratio | 0.63 (0.16) | 0.06 (0.15)

3. Other Pre Specified Outcome: Changes in Anti-growth Hormone Antibody
Time Frame: baseline and 26 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DA-3002 Treatment Group | Non-treatment Control Group
Number analyzed (Participants) | 33 | 31
ng/mL | 0.30 (0.35) | 0.21 (0.54)

ADVERSE EVENTS:
Arm/Group | DA-3002 Treatment Group | Non-treatment Control Group
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/31
Other Adverse Events (participants affected / at risk) | 19/36 | 14/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DA-3002 Treatment Group (N=36) | Non-treatment Control Group (N=31)
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Strabismus correction (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DA-3002 Treatment Group (N=36) | Non-treatment Control Group (N=31)
Enteritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Strabismus correction (Surgical and medical procedures) | 0 | 1
Pyrexia (General disorders) | 5 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No